CLINICAL TRIAL: NCT01601769
Title: Development of a Tissue Sparing Procedure for the Diagnosis and Therapy of Female Precancerous Genital Lesions Combining Endoscopic and Ultrasound Technics.
Brief Title: Tissue Sparing Therapy of Female Precancerous Genital Lesions With VITOM
Acronym: VITOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Giuseppe Vercellino, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOCOLP
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Cervical Preinvasive Disease
Keywords: Cervical preinvasive disease; Colposcopy; Exocolposcopy; Leep
MeSH Terms: interventions — Colposcopy

ARMS (2):
- Colposcopy (Active Comparator): a Carl Zeiss colposcope with a magnification power from 4x to 20x, with green filter.
  Interventions: Device: Colposcopy
- Vitom (Experimental): The VITOM system, consisting of the VITOM scope, xenon light source, HD camera system, AIDA HD documentation system, 1 monitor, and a mechanical support arm (all Karl Storz, Tuttlingen, Germany) is used for video exocolposcopy.
  Interventions: Device: Vitom

INTERVENTIONS:
Device: Vitom — Patients treated and diagnosed by vitom
  Arms: Vitom
Device: Colposcopy — a Carl Zeiss colposcope with a magnification power from 4x to 20x, with green filter.
  Patients treated by colposcopy
  Arms: Colposcopy

SUMMARY:
Object of the study is the evaluation of the use of a rigid laparoscope for the diagnosis and therapy of lesions of the female genital tract as a substitution or a complementary method to colposcopy with the development of new standards for a tissue sparing therapy Use of existing laparoscopic instruments, which allow a better quality level in the diagnosis and therapy than the current routine.

Development of new optics and instruments, which allow a tissue sparing approach Pre and postoperative measurement of the cervical volume, to be sure that the tissue removal is kept to a minimum level Development of qualitaty parameters for the most tissue respecting operations of the uterine cervix Prospective evaluation of the influence of tissue sparing surgery on future pregnancies

ELIGIBILITY:
Inclusion Criteria:

* Karnowsky-Index > 80,
* 18-80 years,
* CIN.

Exclusion Criteria:

* Pregnancy,
* Previous or current cancer,
* Radio therapy of the pelvis,
* Serious internistic accompanying diseases,
* Psychiatric diseases,
* HIV infection,
* Drug addiction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Cervical volume removed | İmmediately after surgery
  Cervical volume removed during the operation is recorded
İntraoperative Complications | During the intraoperative
  Complications encountered during the prodecure
Short term complications | Within 48 hours after operation
  Complications within 48 hours after operation
Late complications | After 48 hours
  Complications occuring after 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Achim Schneider, MD, MPH, Study Director — Charité University Hospital, Berlin, Germany
Locations (1):
- Charité University Hospital, Berlin, State of Berlin, Germany